CLINICAL TRIAL: NCT00645164
Title: Clinical Evaluation of the Photoallergy Potential of Xenaderm Ointment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: H. B. Slade, MD, Healthpoint
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple
Other Study IDs: 011 101 09 002
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Results first posted 2009-04-06 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: wound healing; photoallergenicity; Healthy subjects
MeSH Terms: interventions — Ointments; Granulex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xenaderm (Experimental): Subject serves as own control
  Interventions: Other: Ointment Vehicle; Drug: Xenaderm

INTERVENTIONS:
Other: Ointment Vehicle — Subject acts as own control. 20 mg under Finn chambers
Drug: Xenaderm — 20 mg under Finn chambers

SUMMARY:
The product is being tested to see if exposure to light causes photoallergic reactions on the skin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Stanfield, PhD, Principal Investigator — Suncare Research Laboratories
Locations (1):
- Suncare Research Laboratories, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned: Approximately 60 evaluable subjects. Analyzed: 59 subjects were enrolled in the study, of which 58 were randomized and received test article. 7 subjects were prematurely withdrawn - 1 prior to receiving test articles; 52 subjects completed the study and were evaluable.
Period: Overall Study
Arm/Group | Xenaderm
Started | 59
Completed | 52
Not Completed | 7
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Xenaderm
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 59
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Frequency Distribution of Skin Irritation Scores
Description: Scores based on skin irritation scale of 0 (no reaction) to 7 (large vesiculo-bullous reaction) in whole units. Photoallergic reactions were characterized by irritation scores of 3 or higher.
Time Frame: 48-hours post irradiation
Population: Analysis was based on number of subjects who completed the study.
Measure: Number; unit: Scores on a scale
Arm/Group | Xenaderm
Number analyzed (Participants) | 52
Scores on a scale
  No reaction (0) | 39
  Minimal (doubtful) response (1) | 10
  Definite, mild erythema (2) | 3
  Moderate erythema (3) | 0
  Erythema with slight edema (4) | 0
  Erythema with marked edema (5) | 0
  Erythema w/infiltration w/wo vesiculation (6) | 0
  Large vesiculo-bullous reaction (7) | 0

ADVERSE EVENTS:
Arm/Group | Xenaderm
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Xenaderm
Burning at test site (General disorders) | 3/59 (3)
Itching at test site (General disorders) | 8/59 (8)
Fever (General disorders) | 3/59 (3)
Headache (Nervous system disorders) | 6/59 (6)
Tape reaction (Skin and subcutaneous tissue disorders) | 17/59 (17)

LIMITATIONS AND CAVEATS:
Interpretation of frequency distribution of skin irritation scores was based on long term experience with this type of testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No